CLINICAL TRIAL: NCT06175520
Title: Introduction of Preconception Care Through the Public Health System to Improve Maternal Health and Family Planning Service Utilizations Among Young Women in Rural Bangladesh: A Cluster Randomized Controlled Trial
Brief Title: Introduction of Preconception Care Through Public Health System for Improving MNCH&FP
Acronym: MNCH&FP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Directorate General of Family Planning, Minstry of Health and Family Welfare, Bangladesh (Unknown); Directorate General of Health Services, Minstry of Health and Family Welfare, Bangladesh (Unknown); UNFPA (Unknown); FCDO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: PR-21032
Record Dates: First submitted 2023-11-08; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Feasibility; Acceptability of Health Care
Keywords: Preconception Care; Health System; Maternal Health; Family Planning; Adolescent Pregnancy
MeSH Terms: conditions — Patient Acceptance of Health Care | interventions — Preconception Care

STUDY DESIGN:
Intervention Model Description: Under this model, eligible participants (newlywed married women) from each of the intervention clusters (union catchment area considered as a cluster) will be provided preconception care by community-based healthcare providers. To provide preconception care and counseling the investigators will involve different strategies which include counseling by the Marriage registrar, use of digital platforms to deliver messages, distribution of FP methods, PCC card, and MCH handbook intervention clusters. Overall the intervention components will be evaluated in parallel against a comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preconception care (PCC) intervention (Experimental): There will be 12 clusters under the PCC intervention arm. Eligible participants (newlywed women) in PCC intervention areas will be followed up prospectively. The investigators will enroll around 2,500 participants residing in the study area and with no intention to relocate in the next 2 years. Under this arm, all the relevant healthcare providers and their line managers will be provided training on preconception care. Healthcare providers will enroll the participants using their couple registrars to provide preconception care.
  Interventions: Behavioral: Preconception care (PCC)
- Comparison area (No Intervention): There will be 12 clusters under the comparison arm. Eligible participants will receive services through the existing health system.

INTERVENTIONS:
Behavioral: Preconception care (PCC) — The investigators will introduce PCC through the existing public health system. At the community level facility, healthcare providers will screen the women for some specific health problems and provide necessary supplements. Healthcare providers will screen for health problems such as- infectious diseases (e.g., Tuberculosis), Hypertension, Anaemia, Diabetes Mellitus, Thyroid problems, Sexually Transmitted Infection/Reproductive Tract Infection/Urinary Tract Infection, Nutritional status (e.g., Body mass index), Thalassemia symptoms, Thyroid symptoms, severe Dysmenorrhea, Immunization status, and Symptoms of acute Hepatitis B Virus infection, etc. The provider will also consider age, menstrual history, and reproductive history during preconception screening. If the provider finds any abnormality from the screening test which is a risk for a woman to become pregnant and for her newborn; the woman will be provided proper counseling, treatment, and referral to the appropriate facility.
  Arms: Preconception care (PCC) intervention

SUMMARY:
The goal of this study is to test the feasibility and acceptability of introducing preconception care into the public health system targeting newlywed couples in increasing the uptake of maternal, neonatal health, and family planning services. The Investigators will follow a cluster randomized controlled trial design to implement this study. Twenty-four of the 30 clusters will be selected based on similar characteristics, then will be randomized into intervention and control arms prior to enrollment of the study participants. Therefore, there will be 12 clusters under each arm. Eligible participants from both arms will be surveyed at baseline and 3, 6, 9, 12, 15, 18, 21- and 24-month follow-ups. So, all the newly married couples both in intervention and comparison areas will be followed up prospectively and periodically. The Investigators will introduce preconception care to the existing government health system to ensure healthy pregnancy as well as to improve maternal, child, and adolescent health. For this study, The Investigators propose a package of preconception care interventions such as: screening for nutrition conditions, tobacco use, genetic condition, environmental health, infertility/ sub-fertility, family planning counseling and services, infectious diseases, and Vaccinations.

DETAILED DESCRIPTION:
Bangladesh has one of the world's highest rates of child motherhood. Young motherhood is associated with several risks such as: higher maternal mortality rates, pregnancy complications, and low birth weight babies. A significant proportion of first-time mothers are adolescents and this group of women has a high rate of morbidity and mortality. In Bangladesh, maternity care does not start until the pregnancy is established. The number of births to adolescent mothers has reduced by almost one quarter in the past 18 years but the pace of decline is very slow and adolescent motherhood remains common in rural areas. Preconception care provides an opportunity to optimize the health of potential mothers and to prevent harmful exposures from affecting the developing fetus. In fact, preconception care is the provision of biomedical, behavioral, and social health interventions to women and couples before conception occurs, aimed at improving their health status, and reducing behaviors and individual and environmental factors that could contribute to poor maternal and child health outcomes.

The investigators propose to conduct this study in three Upazilas (Sub-districts) of Gaibandha district in Bangladesh. The sub-districts are: Sundarganj, Palashbari, and Sadullapur. The project will be implemented in collaboration with the Directorate General of Health Services (DGHS) and Directorate General of Family Planning (DGFP).

At the community level, Family Welfare Assistant (FWA) will identify women who want to be pregnant soon (in the next 3 to 6 months) and will send them to FWV at UH&FWC. Our initial target is to identify and enroll newlywed women 6 months prior to pregnancy but at least 3 months will be ensured so that women can get ready to conceive after recovery from any health complications through the preconception screening and treatment procedure. For some health problems, such as infectious diseases like TB, it takes 6 to 9 months to complete the dozes.

FWA maintains a family planning registrar where information of all couples related to use of contraceptives is available. Basically, FWA knows who are using or not using any contraceptive methods, who are pregnant, who are planning for pregnancy and who need what sort of FP methods. From that list they will find those couples and bring them to preconception care from the community level. Apart from FWA, other community-based health workers such as CHCP of Community Clinic and Health Assistant (HA) of DGHS department will also be involved in recruiting the eligible couple under this intervention. Once newlywed couples are identified, they will be referred to UH&FWC for preconception care. If any health problems are diagnosed with those, they will go through proper treatment and newlywed women will be made fit for pregnancy and the other groups may be allowed to go for safe pregnancy. However, at the facility level, healthcare providers especially FWV will provide the preconception care where our main target is to screen the women for some specific health problems and provide necessary supplements. FWV will screen for health problems such as: infectious diseases (e.g., TB), Hypertension, Anaemia, Diabetes Mellitus, Thyroid problems, STI/RTI/UTI, Nutritional status (e.g., BMI), Thalassemia symptoms, Thyroid symptoms, sever Dysmenorrhea, Obesity, Immunization status specially for TT & MR and even Covid-19, and Symptoms of acute HBV infection, etc. Provider will also consider age, menstrual history and reproductive history during preconception screening. Required test for screening these health problems are available at the UH&FWC but for some specific test (like TB test, hemoglobin electrophoresis test) which is not available at FWC, women will be referred to Upazila Health Complex. If provider finds any abnormality from the screening test which is a risk for a woman to become pregnant and for her newborn; woman will be provided proper counseling, treatment, and referral to appropriate Gynae consultants or at facility.

The purpose of preconception care is to rid potential mothers of such health problems even before conception so that she is a healthy individual while carrying her child, which would result in a healthy, developed baby. Preconception care will fulfill this basic right to all potential mothers and ensure the safety of the baby with the help and support of the government health system. The investigators expect the outcome of the intervention is that it will significantly decrease complications during pregnancy and childbirth, adolescent and unintended pregnancies can be prevented to ensure delaying the first births, skilled attendance at ANC, delivery and PNC will be increased, and postpartum family planning practice will be increased to ensure spacing between births. The impact of the project is expected to be healthy pregnancy and birth outcomes and reduced maternal and child morbidity and mortality.

As mentioned, the current system of providing maternal health services starts with pregnancy registration which leaves no opportunity to cure some health complications. Delayed detection of pregnancy and registration with health service providers often cause delay or omit the first ANC which cause different health complications for mother and the newborn. So, the investigator's aim is to avert the health complications by bringing married adolescents to preconception care and remove the risks and make women fit for healthy pregnancy for positive birth outcomes.

Distribution of FP Gift box to the eligible couples: Newlywed couples who are under 20 years of age will be primary target beneficiaries for the first level of intervention. At the onset of intervention, the investigators will provide training to Marriage Registrars (Kazis) on how to counsel newlywed couples and where to refer them for appropriate preconception screening and care. Marriage registrars will be linked with health care providers so that they can work in a team to maximize the outcomes. This will have the added benefit to the midwives, FWVs, FWAs and Kazis establishing a linkage and a working relationship among them.

Delivery of FP Gift box by Marriage Registrar (Kazi), was piloted earlier elsewhere in Bangladesh. In the study area, all the marriage registrars (Kazi) will be involved in this intervention and trained under this study. On the occasions of marriage, marriage registrar will hand over a gift box. Marriage Registrar or Kazi will be sensitized about the importance of family planning specially to delay the first birth of newly married adolescent girls and spacing between births. After the sensitization, a FP gift box will be provided to newlywed couple by Kazi at the time of marriage registration wherever it occurs at Kazi office or at bride's residence homes. FP Gift box contains a comprehensive handbook consist of several information related to husband-wife relationship, relationship with in-laws, food and nutrition, pregnancy plan, access to FP information and services, pregnancy and child care including vaccinations. It covers complete information for continuum of care. Besides, a few Condoms and Pills will be there in the gift box to provide them to newlywed couple so that they can meet their immediate demand just after marriage until they come to contact with family planning worker.

Couple counseling and family engagements: During preconception care and distribution of FP gift FWA, FWV, and MR will arrange couple counselling to involve male partners in the intervention. A training manual will be developed to be used by the health workers and MR for the event of couple counseling. The manual will include the information regarding importance of preconception care, the use of family planning methods, delayed childbearing, spacing between births, skilled care during pregnancy, at child birth, and postnatal period. Besides, the investigators will also incorporate some other important messages related to a healthy lifestyle such: not taking tobacco, not smoking and avoiding passive smoking, husband-wife respectful relationship, consequences of physical and mental violence to pregnant women, foetus, and postpartum women, dental care, physical exercise, healthy diet, etc to ensure healthy pregnancy.

As per the Bangladeshi community context, family members such as husbands, mother-in-law, father-in-law, mother and fathers somehow help and influence young married women in making decision to seek pregnancy-related care. Our intervention will cover the male partners (husbands) in the couple counselling event and other family members especially mother-in-law or mother will be engaged through organizing community events by the health workers. The event like 'Bou-Sasurir Mela' (bride and mother-in-law gathering) will be organized to aware them about the importance of pre-conception care, use of modern family planning methods, delaying adolescent pregnancy and spacing between births.

Digital health intervention using eMIS platform: At the community level, FWA does the eligible couple (ELCO) registration, pregnancy registration, collect information about FP used by the couples, provide FP messages and short-term methods; refer to UH&FWC for LAPM and pregnancy care. The proposed study will take this as an opportunity to use this eMIS platform. The FWA eRegister is an electronic version of the existing paper register. Once an eligible couple is registered, they will be provided with necessary SBCC information related to preconception care as per the design of the program. Targeted client-specific SBCC messages will be developed for the newlywed couples to provide them with family planning and preconception care-related messages.

The adolescent girls women with primi-gravida (first-time young mothers) who are less than 22 years of age in selected Upazillas will be the primary beneficiaries of the second-line intervention. The MCH handbook is one of the tools that have been considered globally to improve access to quality health care by pregnant women including family planning services, ANC, delivery and post-partum services. This is basically an extended version of ANC card that contains information related to ANC, five danger signs, PNC, newborn danger signs, etc. Once a pregnant woman registered by an FWA, she will be provided with MCH Handbook. There is contact number of local midwives in the MCH handbook. Pregnant women will contact to midwife for ANC and follow-up ANC check-ups. MCH hand book keep the track of every information related to ANC, delivery and PNC. Overall, the aim of providing the MCH handbook is to establish a referral linkage between community-based health workers and facility-based healthcare providers to increase the skilled care at antenatal, delivery and postnatal periods including the facility delivery.

Before the intervention, a baseline data collection will be conducted in both the intervention and comparison areas. During the intervention, a regular follow-up will be carried out to collect monitoring data. After the intervention, an end-line data collection will be done to determine the effectiveness of the intervention. However, at baseline and end line, both quantitative and qualitative data collection will be carried out in the intervention, and control Investigators will apply mixed-method approaches to collect data. For performing quantitative analysis, The Investigators use the statistical software package SPSS STATA, or R based on suitability. To analyze the qualitative data of this study, The Investigators will apply the 'Framework Approach'.

ELIGIBILITY:
Inclusion Criteria:

* Newlywed couples who are under 20 years of age

Exclusion Criteria:

-

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2500 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Through baseline and end line questionnaire survey the study will assess the rate of knowledge and practices are increased in terms of modern FP methods among newlywed women | "through study completion, an average of 1 and half years"
  To determine the improvement status of respondent's knowledge and uptake of family planning methods, the investigators anticipating 25% improvement from baseline to end line.
Through baseline and end line questionnaire the study will assess the frequency of pregnancy related complications are reduced | "through study completion, an average of 1 and half years"
  How much pregnancy related complications are reduced will be assessed among the women who received preconception care compared to who did not receive preconception care.
Through baseline and end line questionnaire survey the study will assess the percentage of study participants have proper knowledge about skilled MNCH services | "through study completion, an average of 1 and half years"
  How much knowledge for skilled MNCH care are increased will be measured from among the women who received preconception care and who did not receive preconception care. The investigators are anticipating 25% improvement from baseline to end line
Through baseline and end line questionnaire survey the study will assess the proportion of recently delivered women utilized skilled ANC, DC, and PNC services | "through study completion, an average of 1 and half years"
  To determine the Antenatal care (ANC), Delivery care (DC) and Postnatal care (PNC) uptake by skilled provider, the investigators will follow the criteria of Bangladesh Demographic and Health Survey (BDHS).

SECONDARY OUTCOMES:
Through baseline and end line questionnaire survey the study will assess the rate of delaying first birth among the study participants' | "through study completion, an average of 1 and half years"
  As our study participants are mostly adolescents, preconception care intervention will encourage them to delay their first birth until 20 years of age as per the government guideline. The investigators will assess the delay of first birth among the enrolled women by calculating the time period between their age at enrollment and age at conception within the study period.
Through baseline and end line questionnaire survey the study will assess the rate of unintended pregnancy among the study participants' | "through study completion, an average of 1 and half years"
  To see the status of unintended pregnancy among the adolescents, the investigators will see how many women wanted to have their children at that time in their last pregnancy. The investigators will follow the criteria of BDHS

CONTACTS AND LOCATIONS:
Overall Officials: Bidhan Krishna Sarker, MSS, MPH, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Study data will be jointly owned by icddr,b, and UNFPA. After completion of study activities, summary tables of study results will be available on www.clinicaltrials.gov. After study registration, clinicaltrials.gov provides unrestricted public access to study details including summary tables.
  Study investigators will have access to all participants' data without identifiers. Co-investigators will have access to relevant data as defined in the protocol.
Supporting Information: Study Protocol
Time Frame: After completion of study activities, summary tables of study results will be available on www.clinicaltrials.gov.
Access Criteria: Log in www.clinicaltrials.gov